CLINICAL TRIAL: NCT00344643
Title: A Comparison of 12 Month Daily Wear of Two Novel Hyper-Oxygen Permeable Silicone Hydrogel Contact Lenses (HOP/SiH) and A Control, Standard Oxygen Permeable Lens; and, 30-Night Versus 6-Night Immediate Extended Wear of Two HOP/SiH Lenses.
Brief Title: A Comparison of 12 Month Daily Wear of Two Novel O2 Permeable Silicone Hydrogel CLs (HOP/SiH) and A Control, Standard O2 Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: CIBA VISION (Industry); National Eye Institute (NEI) (NIH)
Responsible Party: H. Dwight Cavanagh, UTSW Medical Center at Dallas
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 0202-112
Record Dates: First submitted 2006-06-23; First posted 2006-06-27 (Estimated); Last update posted 2008-06-23 (Estimated); Status verified 2008-06

CONDITIONS: Contact Lenses, Extended-Wear
Keywords: Comparison of Daily wear versus Extended wear in bacterial binding and corneal epithelial thickness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Silicone Hydrogel Soft Contact Lenses

SUMMARY:
The purpose of this research is to compare the on-eye performance of 12 month daily wear versus 6-night extended wear and 30-night extended wear of novel hyper-oxygen permeable contact lenses by studying its effects on human eyes. Usual and customary care will be given in the form of eyeglasses and/or contact lenses.

DETAILED DESCRIPTION:
The purpose of this research is to compare the on-eye performance of 12 month daily wear versus 6-night extended wear and 30-night extended wear of novel hyper-oxygen permeable contact lenses on bacterial binding to corneal cells and central epithelial thickness. Usual and customary care will be given in the form of eyeglasses and contact lenses. To compare long-term Daily wear vs. immediate Overnight wear (Extended wear) of a new hyper-oxygen permeable silicone hydrogel contact lens on binding of Pseudomonas Aeruginosa to exfoliated human surface corneal cells collected from the eyes of human patients and on central corneal thickness, as follows: 1) a hyper Dk/t lens for 12 months of daily wear, 2) a hyper Dk/t lens for 12 months of de novo 6 night extended wear, and 3) a hyper Dk/t lens for 12 months of de novo 30 night extended wear.

ELIGIBILITY:
Inclusion Criteria: The age requirement for this study is between 18-38 years old. The subject has to have nearsightedness in between -1.00D and -6.00D with regular astigmatism of an amount in both eyes that will not necessitate the need for toric lenses. No prior history of any lens wear within one month of entry into the contact lens phase of the study. Visual acuity of 20/30 or better during test lens wear. Normal anatomy and physiology of the eye. No eye cosmetic use on the day of study visits. Normal appearance of the cornea with slit lamp examination, stable tear film and sufficient tear production. Intraocular pressure less than or equal to 21 mmHg by Goldmann applanation. Absence of any intraocular inflammation. Normal appearance of optic nerve, macula and peripheral retina by direct fundus examination.

Exclusion Criteria: Patients with chronic ocular conditions are excluded from the study (i.e. dry eye, recurrent corneal epithelial erosion). History of allergic eye disease either seasonal or associated with previous contact lens wear. Use of any topically applied ocular medication or systemic medication specifically including but not limited to, antihistamines, aspirin-related drugs, or psychoactive or anti-depressant medication. Oral contraceptives are allowed. Currently suspected or actual pregnancy. Study terminates if pregnancy occurs. Patients will not be enrolled if they are currently in another ophthalmic research project.

Ages: 18 Years to 38 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 187 (Actual)
Dates: Start 2004-10; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Primary - Bacterial binding rates between test articles in both manners of wear - Daily wear and extended wear. | 12 Months

SECONDARY OUTCOMES:
Secondary - Corneal Epithelial thickness measures between test articles in both manners of wear - Daily wear and extended wear. | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Harrison D Cavanagh, M.D., PhD, Principal Investigator — University of Texas, Southwestern Medical Center at Dallas
Locations (1):
- University of Texas Southwestern Medical Center At Dallas, Dallas, Texas, United States

REFERENCES:
- [Derived] Robertson DM, Petroll WM, Cavanagh HD. The effect of nonpreserved care solutions on 12 months of daily and extended silicone hydrogel contact lens wear. Invest Ophthalmol Vis Sci. 2008 Jan;49(1):7-15. doi: 10.1167/iovs.07-0940. PMID 18172068